CLINICAL TRIAL: NCT01726491
Title: Epigenetics and the Origin of Muscle Insulin Resistance in Humans
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Lori R. Roust, Consultant in Endocrinology, Mayo Clinic
Other Study IDs: 11-007028
Record Dates: First submitted 2012-11-08; First posted 2012-11-15 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Diabetes Mellitus Type 2 in Obese; Obesity
Keywords: Insulin resistance; Exercise; Type 2 diabetes mellitus; Obesity; Epigenetic studies
MeSH Terms: conditions — Obesity; Insulin Resistance; Motor Activity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — thigh muscle biopsies bloodsamples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Insulin resistance epigenetics: This experiment will use the Infinium methylation assay to perform epigenome mapping and define patterns of DNA methylation in skeletal muscle and whole blood tissue of metabolically well-characterized lean healthy, obese nondiabetic, and type 2 diabetic volunteers. We will test the hypotheses that
  (1) There is an increased methylation of genes involved in mitochondrial biogenesis and oxidative phosphorylation and altered methylation of promoters of genes coding for extracellular matrix and cytoskeletal proteins in insulin resistance, (2) The altered methylation patterns observed correspond to protein and mRNA expression changes, and (3) There are coordinated patterns of DNA methylation between the skeletal muscle and whole blood tissues in insulin resistance.
- Single bout of exercise: This experiment will test the hypotheses in lean healthy, obese non-diabetic and type 2 diabetic volunteers that
  1. Increased methylation of the PGC-1α promoter predicts a decreased response of this gene to a single bout of exercise, and
  2. Altered methylation of promoters of nuclear encoded mitochondrial genes predicts a decreased response of this gene to a single bout of exercise.
- Eight weeks of exercise: This experiment will test the hypothesis in lean healthy, obese non-diabetic and type 2 diabetic volunteers that
  1. There is decreased methylation of genes involved in mitochondrial biogenesis and oxidative phosphorylation, and the altered methylation corresponds to protein and mRNA (messenger ribonucleic acid) expression changes,
  2. There is altered methylation of genes involved in inflammation and cytoskeletal structure.

SUMMARY:
The investigators are trying to understand the role of DNA (deoxyribonucleic acid) methylation in insulin resistance in skeletal muscle and blood tissues. DNA methylation is a normal chemical process in the body that modifies DNA. By studying this, the investigators hope to better understand the causes of insulin resistance.

DETAILED DESCRIPTION:
Insulin resistance is defined as the decreased ability of insulin to perform its biological function in the muscle, liver and fat. Genetic and environmental factors are known to influence insulin sensitivity. It is not known how this is mediated. This study looks at the role of epigenetics (modifications of proteins associated with DNA and methylation of DNA) in alterations in insulin resistance. We will study lean healthy people, obese non-diabetic people and people with type 2 diabetes to characterize the DNA methylation patterns in muscle in each group. The second aim of the study is to see how a single bout of exercise affects the DNA methylation in the muscle. The third aim looks at the effect of 8 weeks of supervised exercise on the DNA methylation.

ELIGIBILITY:
Volunteers must be:

* 21 - 55 years old
* must be non-lactating, non-pregnant
* not taking medications known to affect glucose or if taking them, on stable doses.
* free of significant heart or lung disease

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Three groups of volunteers will be studied: 1) lean, healthy volunteers, 2)obese volunteers without type 2 diabetes, and 3) volunteers with type 2 diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2012-08; Primary Completion 2016-11-21 (Actual); Study Completion 2016-11-21 (Actual)

PRIMARY OUTCOMES:
DNA methylation of genes in insulin resistance | Baseline to visit 33 (approx 2 months)
  DNA methylation of genes involved in mitochondrial biogenesis, oxidative phosphorylation, extracellular matrix and cytoskeleton proteins in insulin resistance, with an acute episode of exercise, and with eight weeks of training exercise.

SECONDARY OUTCOMES:
mRNA expression of genes | Baseline to visit 33 approx 2 months
  mRNA expression of genes involved in mitochondrial biogenesis, oxidative phosphorylation, extracellular matrix and cytoskeletal signaling are altered in insulin resistance, with an acute episode of exercise and with 8 weeks of exercise training.

CONTACTS AND LOCATIONS:
Overall Officials: Lori Roust, MD, Principal Investigator — Mayo Clinic; Dawn K Coletta, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States